CLINICAL TRIAL: NCT00383539
Title: Lot-to-Lot Consistency Study of the Investigational, Inactivated, Split-Virion Influenza Vaccine in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GID23
Record Dates: First submitted 2006-09-29; First posted 2006-10-03 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Orthomyxoviridae Infection; Influenza; Myxovirus Infection
Keywords: Influenza; Orthomyxoviruses; Inactivated Split-virion influenza vaccine; Adults
MeSH Terms: conditions — Orthomyxoviridae Infections; Influenza, Human | interventions — vaxigrip

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Lot 1
  Interventions: Biological: Inactivated Split-virion influenza vaccine
- 2 (Experimental): Lot 2
  Interventions: Biological: Inactivated Split-virion influenza vaccine
- 3 (Experimental): Lot 3
  Interventions: Biological: Inactivated Split-virion influenza vaccine
- 4 (Active Comparator): Control
  Interventions: Biological: Inactivated Split-virion influenza vaccine

INTERVENTIONS:
Biological: Inactivated Split-virion influenza vaccine — Vaccine Lot 1
  Arms: 1
Biological: Inactivated Split-virion influenza vaccine — Vaccine Lot 2
  Arms: 2
Biological: Inactivated Split-virion influenza vaccine — Vaccine Lot 3
  Arms: 3
Biological: Inactivated Split-virion influenza vaccine — Control Vaccine
  Other Names: Vaxigrip
  Arms: 4

SUMMARY:
The primary objective of this trial is to demonstrate the equivalence, in terms of immunogenicity, of three different industrial lots of the investigational vaccine thereby supporting consistency of the manufacturing process.

Secondary Objectives:

Immunogenicity

To demonstrate that the investigational vaccine induces an immune response at least as good as the one induced by the reference vaccine, in terms of antibody titers.

To assess the immunogenicity of the investigational vaccine using parameters defined in the European Medicines Agency (EMEA) Note for Guidance (CPMP/BWP/214/96).

Safety:

To demonstrate that the investigational vaccine is at least as well tolerated as the reference vaccine, in terms of defined safety profile.

To describe the safety profile after vaccination.

Comfort of the vaccination assessment:

To assess the pain immediately after the injection using a Verbal Rating Scale. To describe the vaccination comfort after the injection using a -Patient-Reported Outcome questionnaire: the Vaccination Comfort Questionnaire.

ELIGIBILITY:
Inclusion Criteria :

* Aged 18 to 60 years on the day of inclusion.
* Informed consent form signed.
* Able to attend all scheduled visits and to comply with all trial procedures.
* For a woman, inability to bear a child or negative urine pregnancy test at the first visit.

Exclusion Criteria :

* Systemic hypersensitivity to egg proteins, chick proteins, or any of the vaccine components, in particular, neomycin, formaldehyde, and octoxinol 9, or history of a life-threatening reaction to the trial vaccine or a vaccine containing the same substances.
* Febrile illness (oral temperature >= 37.5°C, or rectal equivalent temperature >= 38.0°C) on the day of inclusion.
* Participation in another clinical trial in the 4 weeks preceding the trial vaccination.
* Planned participation in another clinical trial during the present trial period.
* Congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroids therapy.
* Unstable chronic illness (defined as illness requiring hospitalization or a clinically significant change in medication in the 12 weeks prior to inclusion) at a stage that could interfere with trial conduct or completion.
* Current abuse of alcohol or drug addiction that may interfere with the subject's ability to comply with trial procedures.
* Blood or blood-derived products received in the past 3 months.
* Any vaccination in the 4 weeks preceding the trial vaccination.
* Vaccination planned in the 4 weeks following the trial vaccination.
* Previous vaccination against influenza (in the previous 6 months).
* Thrombocytopenia or bleeding disorder contraindicating intramuscular vaccination.
* Subject deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized without his/her consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2256 (Actual)
Dates: Start 2006-09; Primary Completion 2007-07 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
To provide information concerning the immunogenicity of an inactivated, split-virion influenza vaccine | 21 Days pot-vaccination

SECONDARY OUTCOMES:
To provide information concerning the safety of an inactivated, split-virion influenza vaccine. | 6 months post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc.
Locations (4):
- Angers, France
- Vilnius, Lithuania
- Madrid, Spain
- Bath, United Kingdom

REFERENCES:
- [Derived] Arnou R, Eavis P, Pardo JR, Ambrozaitis A, Kazek MP, Weber F. Immunogenicity, large scale safety and lot consistency of an intradermal influenza vaccine in adults aged 18-60 years: Randomized, controlled, phase III trial. Hum Vaccin. 2010 Apr;6(4):346-54. doi: 10.4161/hv.6.4.10961. Epub 2010 Apr 15. PMID 20372053
- [Derived] Chevat C, Viala-Danten M, Dias-Barbosa C, Nguyen VH. Development and psychometric validation of a self-administered questionnaire assessing the acceptance of influenza vaccination: the Vaccinees' Perception of Injection (VAPI) questionnaire. Health Qual Life Outcomes. 2009 Mar 4;7:21. doi: 10.1186/1477-7525-7-21. PMID 19261173
- See also: Related Info — http://www.sanofipasteur.com